CLINICAL TRIAL: NCT01863082
Title: Effects of Training in a Heated Pool in Patients With Refractory Hypertension
Brief Title: Resistant Hypertension and Physical Activity Performed in a Heated Pool
Acronym: HAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Edimar Alcides Bocchi, PHD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010/15649-4
Record Dates: First submitted 2013-05-20; First posted 2013-05-27 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Resistant Hypertension
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental): the patients will be submitted to an exercise protocol
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — practice of physical exercise

SUMMARY:
patients with resistant hypertension will be submitted to an exercise protocol in a heated pool for three months

DETAILED DESCRIPTION:
pacient´s blood pressure behavior will be compared before and after intervention

ELIGIBILITY:
Inclusion Criteria:

* patients with uncontrolled blood pressure despite concurrent use of 3 antihypertensive agents, including a diuretic, or the need for more than 3 medications to control blood pressure

Exclusion Criteria:

* poor adherence to the treatment
* obesity
* diabetes
* smokers
* secondary causes of hypertension
* motor disabilities to perform the training

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure value | Change from Baseline in Blood Pressure at 3 months
  participants will be followed for the duration of the exercise protocol, an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lais GB Cruz, Study Chair — Heart Institute (InCor) HC FMUSP; Guilherme V Guimarães, PhD, Principal Investigator — Heart Institute (InCor) HC FMUSP
Locations (1):
- Heart Institute of São Paulo University Medical School, São Paulo, São Paulo, Brazil